CLINICAL TRIAL: NCT05375344
Title: MoVE on Up: Mobility and Voiding Exercises in Older Women With Urinary Incontinence
Brief Title: Mobility and Voiding Exercises in Older Women With Urinary Incontinence (MoVEonUp)
Acronym: MOVEONUP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Uduak Andy, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 849788
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Participants in this group will participate in the home-based exercise group intervention that consists of general balance and strength training, bladder training and urge suppression, and home hazard assessments.
  Interventions: Behavioral: Exercise Group
- Control Group (No Intervention): Participants in this group will receive informational booklets on fall prevention and behavioral treatment for Urgency Incontinence.

INTERVENTIONS:
Behavioral: Exercise Group — Home-based exercise group intervention
  Arms: Exercise Group

SUMMARY:
A prospective, two-arm randomized clinical trial utilizing a multidimensional intervention to reduce falls in older women with Urinary Urge Incontinence. The intervention consist of general balance and strength training, bladder training and urge suppression, and home hazard assessments. The control group will receive informational booklets on fall prevention and behavioral treatment for urinary urge incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 70 or older
* Living independently in the community
* Willingness to be randomized.
* Ability to read and understand English
* Be able to provide informed consent
* Low physical activity (physically active for 30 minutes or more less than or equal to 2 days per week on average over the past 6 months) per PAS
* Ambulatory (defined as patient not confined to bed or wheelchair OR ability to walk with or without an assistive device)
* Self-reported moderate to severe urge-predominant UI based on the ICIQ-SF > 6 (Q 1+2+3)
* Not planning to initiate new UI or overactive bladder (OAB) treatment during the study duration
* Capable of participation in an exercise program without exacerbating any pre-existing condition(s), as determined by the study PI or designee

Exclusion Criteria:

* Pelvic organ prolapse passed the hymen (per patient report)
* Undergoing active treatment for cancer (other than non-melanoma skin cancer)
* Uncorrected visual or hearing loss.
* Other urinary conditions or procedures that may affect continence status for example: urethral diverticulum, previous augmentation cystoplasty
* Progressive neurodegenerative disease e.g. Parkinson's disease, multiple sclerosis per patient report
* History of stroke or carotid sensitivity (i.e. syncopal falls) per patient report
* Unstable cardiac disease per patient report
* Fracture or joint replacement within the last six months per patient report
* Significant cognitive impairment (defined as a modified TICs score of < 27)
* Per PI discretion, participant cannot enroll in study

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in number of falls between the baseline visit and 1 year | 12 months
  number of falls reported in a falls diary

SECONDARY OUTCOMES:
Change in urinary incontinence score on the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) between baseline visit and 1 year | 12 months
  Change in International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF). A minimum score is 0, a maximum score is 21 with a higher score indicating higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Uduak U Andy, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andy UU, Newman DK, Wyman JF, Klusaritz H, Walsh W, Shou H, Koepler N, Schmitz KH, Reaves S, Arya L, Brown RT. The Mobility and Voiding Exercises in Older Women with Urinary Incontinence (MoVEonUp) randomized controlled trial: study protocol and rationale. BMC Geriatr. 2024 Dec 4;24(1):994. doi: 10.1186/s12877-024-05552-7. PMID 39633261